CLINICAL TRIAL: NCT02257112
Title: Measurement of Low-energy Stimulation in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardialen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CL001
Record Dates: First submitted 2014-09-24; First posted 2014-10-06 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multistage low-energy stimulation (Experimental): Multistage low-energy electrical pulses as described in Janardhan AH et al. JACC 2014 Jan7-14:63(1):40-8 will be delivered to a patient in atrial fibrillation. The responses to these stimuli will be recorded.
  Interventions: Device: Multistage low-energy stimulation

INTERVENTIONS:
Device: Multistage low-energy stimulation — The parameters of the Multistage waveform will be altered and the response of the atria will be recorded.

SUMMARY:
Multistage low-energy pulses are being evaluated for their effect on atrial fibrillation during an acute testing procedure.

DETAILED DESCRIPTION:
This is a research feasibility study to evaluate various parameters of the multistage low-energy pulses and their effect on atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* patients indicated for an atrial fibrillation ablation procedure

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of Multistage low-energy pulses to organize, suppress, or terminate atrial fibrillation as determined by changes in atrial fibrillation cycle length, and atrial electrogram morphology. | Patients will be followed during the acute procedure which is expected to average 60 minutes
  Multistage low-energy pulses are delivered to the atria of patients while in atrial fibrillation. The atrial electrograms will be recorded and used to evaluate if there was a change in the atrial fibrillation cycle length, increased organization of the arrhythmia using frequency analysis or if the pulses were able to terminate the atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Haut-Lévêque, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No
No plan to share data. Data has been published in a peer reviewed journal

REFERENCES:
- [Background] Janardhan AH, Gutbrod SR, Li W, Lang D, Schuessler RB, Efimov IR. Multistage electrotherapy delivered through chronically-implanted leads terminates atrial fibrillation with lower energy than a single biphasic shock. J Am Coll Cardiol. 2014 Jan 7-14;63(1):40-8. doi: 10.1016/j.jacc.2013.07.098. Epub 2013 Sep 26. PMID 24076284